CLINICAL TRIAL: NCT03284281
Title: Low-Level Transcutaneous Vagus Stimulation in ST Segment Elevation Myocardial Infarction: TREATMI Study
Brief Title: Low-Level Transcutaneous Vagus Stimulation in ST Segment Elevation Myocardial Infarction: TREAT MI Study
Acronym: TREATMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never initiated; withdrawn prior to receiving IRB approval
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8350
Record Dates: First submitted 2017-08-18; First posted 2017-09-15 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Inflammation
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interventional arm (Experimental): Active TVNS will be performed by use of a Tragus stimulator device with electrodes attached to the tragus of the ear. Stimulator will be applied continuously for 8 hours daily (4 hours twice daily) for 1-week post discharge.
  Interventions: Device: Tragus stimulator
- Control arm (Placebo Comparator): No stimulation will be performed.
  Interventions: Device: Sham Tragus stimulator

INTERVENTIONS:
Device: Tragus stimulator — Tragus nerve stimulation for at least 8 hours per day for 1 week post discharge.
  Arms: Interventional arm
Device: Sham Tragus stimulator — No stimulation will be performed
  Arms: Control arm

SUMMARY:
This study will determine the impact of Transcutaneous Vagus Stimulation(TVNS) and autonomic modulation of inflammation in patients admitted with " acute heart attack."

After admission for "acute heart attack" or "myocardial infarction" patients will be randomized to either TVNS or placebo and their blood samples will be collected at different time points during admission and post discharge.

Blood samples will be analyzed for various markers of inflammation.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

1. Study the effects of TVNS on inflammation in patients with STEMI.
2. Determine the clinical impact of TVNS on 30, 3,6 and 12-month clinical outcomes in patients with STEMI.

B: BACKGROUND AND SIGNIFICANCE:

ST elevation myocardial infarction (STEMI) is the leading cause of death in United States.1 Improved survival following myocardial infarction has largely been due to the contribution of timely reperfusion strategies and advanced pharmacologic management (anti-coagulant and anti-platelet strategies).2 With acute myocardial infarction follows the accompaniment of a systemic and local inflammatory reaction involving both humoral and cell mediated inflammation, which is important in healing and scar formation.3,4 Reperfusion of ischemic myocardium sets the stage for an inflammatory response for the repair and remodeling of the ischemic territory. Experimental evidence has shown that the complement cascade plays an important role in triggering inflammation.3,4 These mechanisms drive the formation of the inflammasome resulting in the release of interleukin (IL)-1 activating expression of inflammatory mediators in necrotic myocardium.5 C-reactive protein (CRP) and IL-6 levels have been shown to correlate to infarction size post-percutaneous coronary intervention.6 Tumor necrosis factor (TNF- α) may be a predominant factor in up regulating the production of IL-6. The presence of significant levels of TNF- α post MI has been shown to correlate to infarct size and recurrent myocardial infarction.4,7 IL-10, an anti-inflammatory marker is important during the late phase of acute inflammation within myocardium in helping to inhibit inflammation while attenuating remodeling, increasing capillary density and improving left ventricular function.8 Expression of TGF-beta isoforms increases in necrotic myocardial regions and may exert anti-inflammatory effects by down regulating proinflammatory cytokine production, chemokine and adhesion molecule synthesis and promoting differentiation of inhibitory lymphocyte subsets. Lastly, TGF- β promotes matrix-stabilizing effects and is key in matrix remodeling and fibrosis in post myocardial infarction tissue and in chronic heart failure.5 Brunetti et. al. outlined the trend in inflammatory biomarkers such as CRP, ESR, and fibrinogen in patients presenting with STEMI receiving fibrinolytic therapy. They reported a peak level of such markers on day 2-3 post-STEMI.9 In a similar study by Brunetti et. al. it was also noted that higher TNF- α levels were associated with subsequent adverse cardiac events.10 Pudil et. al studied the variation in the levels of IL-6, CRP and TNF-alpha among 24 acute myocardial infarction (AMI) patients over 96 hours and determined that IL-6 and TNF- α levels were continually high during the 96 hours, however CRP increased later than IL-6 and peaked at 42 hrs after AMI.11 IL-6 levels seem to be elevated more so in the first 1-3 days following AMI with levels persistently elevated even 3 weeks after AMI.12 Inflammation plays a key role in atherogenesis and several complex interconnected pathways exist that modulate inflammation in STEMI. There remains an intense interest to identify anti-inflammatory therapies that may help reduce the risk of cardiovascular events. A recently published study with an anti-inflammatory agent Losmapimod ( p38 mitogen activated protein kinase), failed to demonstrate any improvement in clinical outcomes.13 It is thought that due to the interplay of several inflammatory cascades, targeting one particular pathway may not provide the desired impact on inflammatory milieu and clinical outcomes.

To the investigator's knowledge, there is no data that suggests that modulating the autonomic nervous system via TVNS (by increasing the parasympathetic tone and reducing the sympathetic nervous system activity) would lead to a reduction in the circulating pro-inflammatory cytokines in patients with STEMI. Since this concept has not been tested previously, the investigators embark on the idea of using autonomic modulation via TVNS to reduce the level of systemic inflammation that is rampant in patients admitted with STEMI.

We hypothesize that:

* TVNS will lead to a reduction in the levels of pro-inflammatory cytokines (such as TNF-α, IL-1, IL-6, CRP, TGF- β) and increase in anti-inflammatory cytokine IL-10, in patients with STEMI. PRIMARY HYPOTHESIS
* TVNS may lead to a reduction in clinical adverse events (assessed cumulatively over a period of one-year post-STEMI). Major Adverse Cardiac Events- death, myocardial infarction, heart failure, readmission for acute coronary syndrome or heart failure, repeat revascularization. SECONDARY HYPOTHESIS

C: PRELIMINARY STUDIES:

The investigators intend to perform a pilot study to:

* Determine the anti-inflammatory effect of TVNS in patients with STEMI.
* Determine the impact of TNS on adverse clinical events post-STEMI.

D: RESEARCH DESIGN AND METHODS:

Design: Prospective study

Intended sample size: 50

Patients will be recruited from the inpatient services of OUHSC.

After full written informed consent be randomly assigned (1:1) to active TVNS vs. control group with no TNS. The patients will be requested to refrain from discussing the details of their treatment with other patients in the hospital and with the physicians, nurses and the rest of clinic staff. The clinical coordinator who will not participate in any of the other study related assessments will instruct the patients on the proper use of the device. These study personnel will be designated to address the patients' questions and concerns as well as to record any side effects related to the use of the device.

Active TVNS will be performed by use of a transcutaneous electrical nerve stimulation 14 device with electrodes attached to the tragus of the ear, which is innervated by an auricular branch of the vagus nerve. The SALUSTIM Digital TENS Unit, distributed within the US by US Medical Inc. will be used for TVNS or sham stimulation. The device will be connected to a clip electrode that will be attached to the external ear. In the active group, the ear clip electrode will be attached to tragus in the active stimulation group (Figure 3). The ear clip electrode has not been previously reviewed by the FDA for purposes such as this but has been classified as a non-significant risk device per FDA guidelines. It has been however studied in Europe and is available in the European market under the name SaluSTIM®. The TENS unit will be set at a pulse width of 100 μs and a pulse frequency of 20 Hz. Amplitude will be titrated to the level of sensory threshold, typically in the range of 10-50 mA. The stimulation strength will be gradually increased until the patient experiences mild discomfort, and then decreased by 1 mA below that threshold. TENS will be applied continuously for 8 hours daily (4 hours twice daily) for 1 week.

During index hospitalization: The patients randomized to TVNS will be stimulated soon after the consent is obtained. The initial stimulation duration will be for 4 hours. After this, the patients will follow the stimulation times of 6AM-10AM and 5PM-9PM.

Post discharge: Patients will be instructed to apply the devices at the same time each day for 1 week to avoid discrepancy in the time of stimulation. The optimal timing will be 7AM-11 AM and 5 PM- 9 PM. However, the patients will be given a window of 5AM-Noon(7 hours) and 4PM-11PM( 7 hours) and will be told to use the unit for 4 hours continuously during this window. The clinical coordinator will instruct the patients on the proper use of the device. The choice of treatment for STEMI will be left at the discretion of the treating physician.

During the baseline hospital admission, a complete history and physical examination will be done by one of the research co-ordinators. Laboratory data, electrocardiographic data, and echocardiographic data will also be reviewed. 10ml of blood will be drawn for cytokine analysis.

Baseline sample: a 10 ml blood sample will be collected upon arrival and prior to angioplasty/stenting. This could be performed either in the emergency room or in the catheterization laboratory after informed consent obtained.

Subsequent sample collection: a 10 ml blood sample will be collected 12, 24 and 48 hours post PCI.

Follow up sample: a 10 ml blood sample will be drawn a week and a month after discharge during a regular clinic visit.

Sample analysis: Samples will be collected in BD red top glass tube. The tube will be left in a standing position for about 30-45 minutes and then centrifuged at room temperature, 1500g for 10 minutes. Serum will be removed immediately and frozen in 0.5 cc aliquots at -80C. The samples (in blocks) will then be transferred to OU Medical Center/Research lab where levels of CRP, TNF- α, IL-1, IL-6, IL-10 and TGF- β will be measured in batches.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18 years or older) with ST Segment elevation myocardial infarction (STEMI) undergoing primary PCI.

Exclusion Criteria:

* Patients transferred in from outside facilities after having received fibrinolytic therapy
* patients in cardiogenic shock
* patients with pacemakers and defibrillators
* patients undergoing urgent coronary bypass surgery
* cardiac arrest patients
* mechanical complications (ventricular septal defects, acute papillary muscle rupture, free wall rupture)
* patients on mechanical ventilation
* chronic inflammatory disease (systemic lupus erythematosus, rheumatoid arthritis, and Crohn's disease), or receiving therapy with steroids, cyclosporine, or methotrexate
* unilateral or bilateral vagotomy
* pregnant patients
* prisoners
* end stage renal disease on dialysis
* history of recurrent vasovagal syncope, Sick sinus syndrome, 2nd or 3rd degree AV block.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Change in CRP levels | Change from admission to 1 month post discharge
  mg/dL
Change in TNF-alpha and TGF-beta levels | Change from admission to 1 month post discharge
  ng/L
Change in interleukin levels (IL-1,IL-6,IL-10) | Change from admission to 1 month post discharge
  ng/L

SECONDARY OUTCOMES:
Major adverse cardiac events | Admission to 1 year post discharge
  Death,MI,Stroke,repeat revascularization,Heart failure related admission

CONTACTS AND LOCATIONS:
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided